CLINICAL TRIAL: NCT02555566
Title: Role of Epoxyeicosatrienoic Acids in Chronic Allograft Nephropathy
Brief Title: Role of Epoxyeicosatrienoic Acids in Chronic Allograft Nephropathy - The TRANSPLANT-EETs Study
Acronym: TRANSPLANTEETs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2013/150/HP
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Kidney Transplant Recipients
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kidney transplant recipients (Experimental): blood sampling is done for determination of EPHX Lys55Arg and other polymorphisms status in Kidney transplant recipients.
  flow-mediated distal stimulation of the forearm radial artery by cutaneous heating is assessed for evaluation of EEts level in Kidney transplant recipients.
  Interventions: Procedure: Blood sampling; Procedure: flow-mediated distal stimulation of the forearm radial artery by cutaneous heating

INTERVENTIONS:
Procedure: Blood sampling — Blood sampling is done for Kidney transplant recipients for evaluation of the polymorphisms and EETs dosage
Procedure: flow-mediated distal stimulation of the forearm radial artery by cutaneous heating — Flow-mediated distal stimulation of the forearm radial artery by cutaneous heating for Kidney transplant recipients

SUMMARY:
Endothelial lesions within the transplanted kidney are a major determinant of chronic allograft nephropathy. Epoxyeicosatrienoic acids (EETs) are endothelium-derived hyperpolarizing factors with anti-inflammatory, antiproliferative and vasodilator properties.

The main goal of the investigators' study is to evaluate whether genetic polymorphisms of specific enzymes responsible for the bioavailability of EETs are associated with post-transplant kidney function.

To this end, 80 kidney transplant recipients will be included. Prespecified genetic polymorphisms of CYP 2J2, CYP 2C8, CYP 2C9, CYP 2C9, CYP 2C19 and EPHX2 will be determined. Kidney function will be recorded 3, 6, 12 and 36 months after transplantation. Flow-mediated dilatation, EETs and circulating biomarkers of endothelial function will be measured in the radial artery.

The expected results of this study to provide preliminary evidence supporting a beneficial role of an increase in the bioavailability of EETs in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 75 yo
* Caucasian (because of different CYP epoxygenase polymorphisms)
* First kidney transplantation performed in Rouen University Hospital after 2000, and at least 12 months before inclusion
* Patient having read, understood and approved the informed consent
* Efficient contraception in child-bearing aged women
* Regular health insurance

Exclusion Criteria:

* Primary non-function, or allograft loss before 1 year
* Previous kidney transplantation
* History of psychiatric, psychologic or sensorial disorder preventing the patient from correctly understanding the protocol
* History of bilateral arm or forearm arteriovenous fistula
* Counter-indication to trinitrin
* Insufficient understanding of written or spoken French language
* Liberty-deprived patient
* Pregnancy or absence of contraception in child-bearing aged women
* Patient enrolled in another research protocol within 2 weeks before inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Difference between patients with the EPHX2 Lys55Arg polymorphism and patients without in estimated Glomerular Filtration Rate (eGFR) | 12 Months after transplantation
  eGFR Scores range from 0 [kidney failure] to >90 [normal function]

SECONDARY OUTCOMES:
Difference between patients with the EPHX2 Lys55Arg polymorphism and patients without in estimated Glomerular Filtration Rate (eGFR) | 3 Months after transplantation
  eGFR Scores range from 0 [kidney failure] to >90 [normal function]
Difference between patients with the EPHX2 Lys55Arg polymorphism and patients without in estimated Glomerular Filtration Rate (eGFR) | 6 Months after transplantation
  eGFR Scores range from 0 [kidney failure] to >90 [normal function]
Difference between patients with the EPHX2 Lys55Arg polymorphism and patients without in estimated Glomerular Filtration Rate (eGFR) | 36 Months after transplantation
  eGFR Scores range from 0 [kidney failure] to >90 [normal function]
Difference between patients with specified polymorphisms and patients without in estimated Glomerular Filtration Rate (eGFR) | 3 Months after transplantation
  eGFR Scores range from 0 [kidney failure] to >90 [normal function]
Difference between patients with specified polymorphisms and patients without in estimated Glomerular Filtration Rate (eGFR) | 6 Months after transplantation
  eGFR Scores range from 0 [kidney failure] to >90 [normal function]
Difference between patients with specified polymorphisms and patients without in estimated Glomerular Filtration Rate (eGFR) | 12 Months after transplantation
  eGFR Scores range from 0 [kidney failure] to >90 [normal function]
Difference between patients with specified polymorphisms and patients without in estimated Glomerular Filtration Rate (eGFR) | 36 Months after transplantation
  eGFR Scores range from 0 [kidney failure] to >90 [normal function]
Difference between blood EETs concentration at baseline and after distal cutaneous heating for patients with the specified polymorphisms. | Day 1
  EEts plasma concentration is measured using liquid chromatography coupled to tandem mass spectrometry before and after distal cutaneous heating. Unit is ng per mL
Difference between blood EETs concentration at baseline and after distal cutaneous heating for patients without the specified polymorphisms. | Day 1
  EEts plasma concentration is measured using liquid chromatography coupled to tandem mass spectrometry before and after distal cutaneous heating. Unit is ng per mL
Difference between variation of diameter of the forearm radial artery after distal cutaneous heating for patients with the specified polymorphisms. | Day 1
  Variation of diameter of the radial artery is measured in millimeter.
Difference between variation of diameter of the forearm radial artery after distal cutaneous heating for patients without the specified polymorphisms. | Day 1
  Variation of diameter of the radial artery is measured in millimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique GUERROT, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France